CLINICAL TRIAL: NCT03292315
Title: The Efficacy of a Once Weekly Glucagon-Like Peptide-1 Agonist on Body Weight/Composition and Metabolic Parameters in Persons With SCI
Brief Title: Once Weekly GLP-1 in Persons With Spinal Cord Injury
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Director, Clinical Investigator, National Center for the Medical Consequences of Spinal Cord Injury, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAU-17-038
Record Dates: First submitted 2017-09-20; First posted 2017-09-25 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Spinal Cord Injuries; Insulin Resistance; Pre Diabetes; Obesity
Keywords: Glucagon-Like Peptide-1
MeSH Terms: conditions — Spinal Cord Injuries; Insulin Resistance; Glucose Intolerance; Obesity | interventions — semaglutide; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Semaglutide 1MG Injection [Ozempic] (Experimental): 20 subjects will be randomized to receive once weekly injection of Semaglutide (Ozempic1mg) for 26 weeks.
  Interventions: Drug: Semaglutide 1MG Injection [Ozempic]
- No Intervention (Other): 10 subjects will be randomized to receive no intervention for 26 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Drug: Semaglutide 1MG Injection [Ozempic] — Once weekly injection of 1mg of Semaglutide.
  Arms: Semaglutide 1MG Injection [Ozempic]
Other: No Intervention — No injection will be administered
  Arms: No Intervention

SUMMARY:
Chronic spinal cord injury (SCI) results in adverse soft tissue body composition changes and an extremely sedentary lifestyle. These abrupt changes often lead to a high prevalence of cardiometabolic diseases, such as impaired glucose tolerance/diabetes mellitus and dyslipidemia, conditions which predispose those with SCI to an increased risk for cardiovascular disease compared to the general population. Due to paralysis and wheel chair dependence, maintaining an adequate level of physical activity to counteract these deleterious metabolic changes presents a unique obstacle because conventional first line interventions are lifestyle modifications (e.g., diet and exercise), which may be difficult to achieve. Recently, a new medication has been approved by the Food and Drug Administration to improve glycemic control in individuals with diabetes mellitus, and it has also been investigated as an off-label treatment to induce weight loss. Glucagon-like peptide-1 (GLP-1) agonists are a class of drugs designed to mimic the endogenous incretin hormones released from the gut in a glucose dependent manner following a meal. The mechanisms of action for this drug class of medications include stimulation of glucose-dependent insulin secretion, inhibiting glucagon release, slowed gastric emptying, and reduction of postprandial glucose excursions following food intake. In addition to improved glycemic control, this class of medications also shows promise for its non-glycemic action of facilitating weight loss. The method of delivery of the GLP-1's is by self-administered injections once daily or once weekly, depending on the severity of the clinical case and therapeutic targets for a specific patient.

DETAILED DESCRIPTION:
Obesity is an underlying condition that predisposes to the development of several medical disorders and diseases. It is well appreciated that obesity has reached pandemic proportions in Western societies. The World Health Organization (WHO) estimates that 1.9 billion adults worldwide are overweight and 600 million of these individuals are further sub-classified as obese, with a 44% estimated burden for type 2 diabetes mellitus (T2DM) being attributed to being overweight/obese, as well as a 23% estimated burden for heart disease ("Obesity and overweight," 2016). Excess adipose tissue is assumed to play an integral role in the pathogenesis of vascular dysfunction and the development of T2DM (Lau, Dhillon, Yan, Szmitko, & Verma, 2005).

During the acute and chronic phases of SCI, marked adverse changes occur in soft tissue body composition and associated carbohydrate and lipid metabolism. After an initial rapid loss of lean tissue below the neurological level of injury, a more insidious and progressive lean tissue loss is observed (Modlesky et al., 2004; Spungen et al., 2003), which is accompanied by an increased total body adiposity (Spungen et al., 2003), with accumulation of fat in the abdominal (e.g., visceral) compartment (Gorgey, Mather, Poarch, & Gater, 2011). These adverse changes to body composition contribute to, and are associated with, a higher prevalence of insulin resistance and disorders of carbohydrate metabolism (e.g., impaired glucose tolerance and T2DM) than that reported in the general population (Bauman & Spungen, 1994). The primary approach to treat T2DM in the general population is diet and exercise (i.e., lifestyle modification). Of note, the profound inactivity and adverse soft tissue body composition changes that occur in individuals after SCI result in metabolic morbidity which is extremely difficult to manage with lifestyle modification alone. Conventional therapeutic strategies employed in the adjunctive treatment of carbohydrate metabolism disorders in the general population include several pharmacological approaches to maintain and improve glycemic control are in standard practice and include reducing the serum glucose concentration (i.e., insulin, sulphonylureas, thiazolidinediones or glitazones), suppressing hepatic gluconeogenesis (i.e., insulin, biguanides), stimulating endogenous insulin secretion (i.e., sulphonylureas), and/or by inhibiting glucose renal reabsorption and increasing glycosuria (i.e., SGLT-2 inhibitors).

In 2005 a new class of drugs was approved for the treatment for T2DM by targeting the GLP-1 receptor. Exenatide is a GLP-1 agonist that acts as an incretin hormone, and it belongs to a class of gastrointestinal hormones which are released from the L cells of the intestines in response to food ingestion that, as one of its mechanisms of action, increase insulin secretion from pancreatic beta cells (Vilsboll et al., 2003). This phenomenon that was coined "the incretin effect" in the 1960's described the significantly higher plasma insulin levels following orally versus intravenously administered glucose, which can account for 50 to 70% of the insulin secretion observed after food intake (Baggio & Drucker, 2007). Treatment with GLP-1's has increased over the past several years because of their mechanism of action to increase insulin secretion, inhibit glucagon release in a glucose-dependent manner, thus minimizing the risk for hypoglycemia (Baggio & Drucker, 2007; Nauck, Stockmann, Ebert, & Creutzfeldt, 1986; Vilsboll, Krarup, Madsbad, & Holst, 2002). Numerous multi-ethnic and multi-national trials have been performed with exenatide, but none have been reported in persons with SCI. Previous investigation with exenatide once-weekly in able-bodied individuals has resulted in weight loss ranging from 1.6 to 3.9 kg following 24 weeks of intervention (Bergenstal et al., 2010; Blevins et al., 2011; Buse et al., 2013; Chiquette, Toth, Ramirez, Cobble, & Chilton, 2012; Davies et al., 2013; Diamant et al., 2010; Drucker et al., 2008; Inagaki, Atsumi, Oura, Saito, & Imaoka, 2012; Ji et al., 2013; Russell-Jones et al., 2012). As such, to date there is no evidence of the potential efficacy of exenatide to result in weight loss, improve glycemic control, and/or reduce insulin resistance in persons with SCI.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age 18 to 69;
2. Chronic (e.g., duration of injury greater than 3 years) stable SCI (regardless of level of neurological injury);
3. ASIA A-D (non-ambulatory defined as not able to weight bear for more than 20% of the day);
4. Obese Percent Body Fat defined as > 25% for men and > 35% for women (as determined by screening DXA scan);
5. Insulin Resistant as determined at screening: (FPI, ≥15 µU/ml); -OR-
6. Pre-diabetic, as determined by any one of the following:

   1. HbA1C ≥ 5.7% and < 6.4%; or
   2. Impaired glucose tolerance by FSG ≥100 mg/dl and < 125 mg/dl and/or the 2 hour serum glucose concentration (after an OGTT) ≥ 140 mg/dl and < 200 mg/dl

Exclusion Criteria:

1. Personal history of or family history of medullary thyroid carcinoma;
2. History of multiple endocrine neoplasia syndrome type 2;
3. History of pancreatitis;
4. Existing diagnosis of diabetes mellitus, or the results from screening OGTT that identify diabetes mellitus (previously undiagnosed); laboratory thresholds for exclusion will be as follows: HbA1C ≥6.5%, fasting plasma glucose >126 mg/dl, or 2 hour value >200 mg/dl;
5. Receiving treatment for impaired glucose metabolism (i.e., insulin, secretagogues, or other agents to modify peripheral insulin sensitivity or serum glucose concentration);
6. Reduced kidney function (by glomerular filtration rate (GFR <60 ml/min) or liver function tests (any single LFT ≥ 2.5 times above the upper limit of normal) as determined by test results at screening and any time point of the study;
7. Elevated calcitonin level (as determined at screening to rule out thyroid cancer);
8. Pregnancy or women who may become pregnant during the course of the study, or those who are nursing;
9. Medically unstable;
10. Acute illness or infection;
11. Diminished mental capacity; and
12. Inability or unwillingness of subject to provide informed consent.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Body Weight | Baseline, Week 13, Week 26
  Efficacy of GLP-1 to reduce total body weight determined by Dual Energy Absorptiometry (DXA)
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | Baseline, Week 13, Week 26
  Efficacy of GLP-1 to reduce HOMA-IR
Homeostatic Model Assessment of Beta-Cell Function (HOMA-B) | Baseline, Week 13, Week 26
  Efficacy of GLP-1 to increase HOMA-B

SECONDARY OUTCOMES:
Body Fat | Baseline, Week 13, Week 26
  Efficacy of GLP-1 to reduce total body fat determined by Dual Energy Absorptiometry (DXA)
Glycated Hemoglobin (HbA1C) | Baseline, Week 13, Week 26
  Efficacy of GLP-1 to reduce HbA1C

CONTACTS AND LOCATIONS:
Locations (1):
- Kessler Institute for Rehabilitation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cirnigliaro CM, La Fountaine MF, Sauer SJ, Cross GT, Kirshblum SC, Bauman WA. Preliminary observations on the administration of a glucagon-like peptide-1 receptor agonist on body weight and select carbohydrate endpoints in persons with spinal cord injury: A controlled case series. J Spinal Cord Med. 2024 Jul;47(4):597-604. doi: 10.1080/10790268.2023.2207064. Epub 2023 May 9. PMID 37158751